CLINICAL TRIAL: NCT06901180
Title: Evaluation of Short Scar Periareolar Inferior Pedicle Reduction Mammoplasty in Oncoplastic Breast Surgery
Brief Title: in Our Study we Compare Results of Two Oncoplastic Breast Surgery (Short Scar Reduction Mammoplasty and Wise Pattern Reduction Mammoplasty) as Surgical Treatment of Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Gadelkarim Mohamed, asistant lecturer, Sohag University
Other Study IDs: soh-med-25-3-2md
Record Dates: First submitted 2025-03-17; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Evaluation of Short Scar Periareolar Inferior Pedicle Reduction Mammoplasty in Oncoplastic Breast Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- short scar periareolar inferior pedicle reduction mammoplasty: oncoplastic reduction mammoplasty through peri-areolar incision
  Interventions: Procedure: short scar periareolar inferior pedicle reduction mammoplasty
- wise pattern reduction mammoplasty: reduction mammoplasty through inverted T incision

INTERVENTIONS:
Procedure: short scar periareolar inferior pedicle reduction mammoplasty — reduction mammoplasty that minimizes scar with better cosmetic outcomes
  Groups: short scar periareolar inferior pedicle reduction mammoplasty

SUMMARY:
in our study we compare results of two oncoplastic breast surgery (short scar reduction mammoplasty and wise pattern reduction mammoplasty) as surgical treatment of breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with ages ranging from 25 to 75 years.
2. Patients with operable breast cancer (Stage I, II and IIIa).
3. Patients with moderate to large /ptotic breasts.

Exclusion Criteria:

1. Patients with a contraindication to breast conservative surgery:

   1. Multi-centric disease that can't be incorporated by local excision through a single incision that achieves adequate safety margin and satisfactory cosmetic results.
   2. inflammatory carcinoma.
   3. Contraindications to postoperative radiation e.g. pregnancy, pre-existing lung disease with reduced diffusing capacity and pulmonary TB.
   4. diffuse suspicious malignant micro-calcification on mammography.
   5. inability to attain negative surgical margins.
   6. cardiomyopathy
   7. connective tissue disorders with significant vasculitis.
2. Previous chest wall or breast radiation.
3. Patients' refusal participation.

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female patients aged from 25 years to 75 years with early breast cancer that meet inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
oncological outcomes | 1 year
  detect incidence of local recurrence of malignancy
post operative complications | 1 month
  surgical complications
cosmetic outcomes | 1 year
  patients' satisfaction with their breast

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Sohag Governorate, Egypt